CLINICAL TRIAL: NCT03049878
Title: Efficacy of Preoperative Administration of Paracetamol-codeine on Pain Following Impacted Mandibular Third Molar Surgery: a Randomized, Split-mouth, Placebo-controller, Double-blind Clinical Trial
Brief Title: Efficacy of Preoperative Administration of Paracetamol-codeine on Pain Following Impacted Mandibular Third Molar Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Maria Paola Cristalli, DDS PhD, Clinical Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2704/21.02.2013
Record Dates: First submitted 2017-01-24; First posted 2017-02-10 (Actual); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: To Control Pain After Third Molar Surgery
Keywords: postoperative pain; paracetamol; codeine; tooth extractions; analgesia; premedication
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — acetaminophen, codeine drug combination

STUDY DESIGN:
Intervention Model Description: A randomized, split-mouth, placebo-controlled, double-blind clinical trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- analgesic group (Active Comparator): preoperative oral dose of paracetamol-codeine
  Interventions: Drug: Paracetamol Codeine
- placebo group (Placebo Comparator): preoperative placebo (starch)
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Paracetamol Codeine — preoperative administration
  Arms: analgesic group
Drug: Placebo Oral Tablet — preoperative administration
  Arms: placebo group

SUMMARY:
Objectives:

The aim of this study was to determine the effectiveness of preoperative administration of single-dose of paracetamol-codeine, in the relieving of acute post-operative pain after the surgical removal of an impacted mandibular third molar.

Materials and Methods:

The study cohort consisted of 32 Caucasian outpatients, giving a total of 64 bilateral symmetrical impacted mandibles. Patients were randomized in two experimental groups to receive a preoperative oral dose of paracetamol-codeine (analgesic group) or a placebo (placebo group) at the first and second surgeries. Study participants were asked to record pain intensity scores during the operation and the next 2 days, the time of the first request for rescue analgesic, and the total number of postoperative-supplement paracetamol-codeine tablets.

ELIGIBILITY:
Inclusion Criteria:

* absence of systemic pathologies (ASA class I);
* non-smoker;
* not pregnant or lactating;
* good oral hygiene;
* no drug consumption for 10 days before the operation;
* bilateral impacted mandibular third molars with comparable position, depth and inclination;
* presence of the first and second molars;
* absence of painful symptoms and associated inflammatory or osteolytic pathologies in a radiographic examination;
* extraction difficulty index of >7 according to Pederson's scale and a degree of IV (complex procedures) on a modified version of Parant's scale.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-02-21 (Actual); Primary Completion 2015-09-20 (Actual); Study Completion 2016-09-10 (Actual)

PRIMARY OUTCOMES:
Pain measurement assessed with the Numerical Rating Scale-11 (NRS-11) during the operative day. | All study participants were asked to record the pain intensity score at 1:00 pm during the operative day
  The primary outcome of the study was the post-operative pain. Before surgery, patients were instructed to complete the Numerical Rating Scale-11 (NRS-11), which consisted of an interval scale ranging from 0 ("no pain") to 10 ("maximum pain")
Pain measurement assessed with the Numerical Rating Scale-11 (NRS-11) during the operative day. | All study participants were asked to record the pain intensity score at 6:00 pm during the operative day
  The primary outcome of the study was the post-operative pain. Before surgery, patients were instructed to complete the Numerical Rating Scale-11 (NRS-11), which consisted of an interval scale ranging from 0 ("no pain") to 10 ("maximum pain")
Pain measurement assessed with the Numerical Rating Scale-11 (NRS-11) during the operative day. | All study participants were asked to record the pain intensity score at 11:00 pm during the operative day
  The primary outcome of the study was the post-operative pain. Before surgery, patients were instructed to complete the Numerical Rating Scale-11 (NRS-11), which consisted of an interval scale ranging from 0 ("no pain") to 10 ("maximum pain")
Pain measurement assessed with the Numerical Rating Scale-11 (NRS-11) during the 2th day after surgery. | All study participants were asked to record the pain intensity score at 8:00 am during the 2th day after surgery
  The primary outcome of the study was the post-operative pain. Before surgery, patients were instructed to complete the Numerical Rating Scale-11 (NRS-11), which consisted of an interval scale ranging from 0 ("no pain") to 10 ("maximum pain")
Pain measurement assessed with the Numerical Rating Scale-11 (NRS-11) during the 2th day after surgery. | All study participants were asked to record the pain intensity score at 1:00 pm during the 2th day after surgery
  The primary outcome of the study was the post-operative pain. Before surgery, patients were instructed to complete the Numerical Rating Scale-11 (NRS-11), which consisted of an interval scale ranging from 0 ("no pain") to 10 ("maximum pain")
Pain measurement assessed with the Numerical Rating Scale-11 (NRS-11) during the 2th day after surgery. | All study participants were asked to record the pain intensity score at 6:00 pm during the 2th day after surgery
  The primary outcome of the study was the post-operative pain. Before surgery, patients were instructed to complete the Numerical Rating Scale-11 (NRS-11), which consisted of an interval scale ranging from 0 ("no pain") to 10 ("maximum pain")
Pain measurement assessed with the Numerical Rating Scale-11 (NRS-11) during the 2th day after surgery. | All study participants were asked to record the pain intensity score at 11:00 pm during the 2th day after surgery
  The primary outcome of the study was the post-operative pain. Before surgery, patients were instructed to complete the Numerical Rating Scale-11 (NRS-11), which consisted of an interval scale ranging from 0 ("no pain") to 10 ("maximum pain")
Pain measurement assessed with the Numerical Rating Scale-11 (NRS-11) during the 3th day after surgery. | All study participants were asked to record the pain intensity score at 8:00 am during the 3th day after surgery
  The primary outcome of the study was the post-operative pain. Before surgery, patients were instructed to complete the Numerical Rating Scale-11 (NRS-11), which consisted of an interval scale ranging from 0 ("no pain") to 10 ("maximum pain")
Pain measurement assessed with the Numerical Rating Scale-11 (NRS-11) during the 3th day after surgery. | All study participants were asked to record the pain intensity score at 1:00 pm during the 3th day after surgery
  The primary outcome of the study was the post-operative pain. Before surgery, patients were instructed to complete the Numerical Rating Scale-11 (NRS-11), which consisted of an interval scale ranging from 0 ("no pain") to 10 ("maximum pain")
Pain measurement assessed with the Numerical Rating Scale-11 (NRS-11) during the 3th day after surgery. | All study participants were asked to record the pain intensity score at 6:00 pm during the 3th day after surgery
  The primary outcome of the study was the post-operative pain. Before surgery, patients were instructed to complete the Numerical Rating Scale-11 (NRS-11), which consisted of an interval scale ranging from 0 ("no pain") to 10 ("maximum pain")
Pain measurement assessed with the Numerical Rating Scale-11 (NRS-11) during the 3th day after surgery. | All study participants were asked to record the pain intensity score at 11:00 pm during the 3th day after surgery
  The primary outcome of the study was the post-operative pain. Before surgery, patients were instructed to complete the Numerical Rating Scale-11 (NRS-11), which consisted of an interval scale ranging from 0 ("no pain") to 10 ("maximum pain")

OTHER OUTCOMES:
Number of patients using rescue therapy | Number of patients using rescue therapy on the same day from the end of the surgery and during 2 days after operative days
  Number of patients using rescue therapy during 3 days after surgery
Time of analgesic medication | Time elapsed from the end of surgery until the first intake of analgesic medication on the same day of the surgery
  Time elapsed from the end of surgery until the first intake of analgesic medication (minutes)
Number of paracetamol-codeine tablets | Number of paracetamol-codeine tablets taken by the patients during the 3 days after surgery
  Total number of paracetamol-codeine tablets with the same formulation taken by the patient in relation to the pain symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Maria Paola Cristalli, DDS, Principal Investigator — University of Roma La Sapienza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cristalli MP, La Monaca G, De Angelis C, Pranno N, Annibali S. Efficacy of Preoperative Administration of Paracetamol-Codeine on Pain following Impacted Mandibular Third Molar Surgery: A Randomized, Split-Mouth, Placebo-Controlled, Double-Blind Clinical Trial. Pain Res Manag. 2017;2017:9246352. doi: 10.1155/2017/9246352. Epub 2017 Feb 23. PMID 28325960